CLINICAL TRIAL: NCT04817241
Title: Clinical Evaluation of ASTX727 in Combination With Venetoclax All-Oral Therapy vs Standard of Care Cytarabine and Anthracycline Induction Chemotherapy for Younger FLT3WT Patients With ELN High- Risk Acute Myeloid Leukemia
Brief Title: Testing Oral Decitabine and Cedazuridine (ASTX727) in Combination With Venetoclax for Higher-Risk Acute Myeloid Leukemia Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-02246; NCI-2021-02246 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICCNCIHEM10417; 10417 (Other: Yale University Cancer Center LAO); 10417 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; Cytarabine; Daunorubicin; decitabine and cedazuridine drug combination; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (decitabine and cedazuridine, venetoclax) (Experimental): Patients receive ASTX727 PO QD at the recommended phase II dose and venetoclax PO QD on days 1-28 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Decitabine and Cedazuridine; Drug: Venetoclax
- Arm II (cytarabine, daunorubicin) (Active Comparator): Patients receive cytarabine IV over 24 hours on days 1-7 of each cycle and daunorubicin IV over 10-30 minutes on days 1-3 of each cycle. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy throughout the trial.
  Interventions: Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cytarabine; Drug: Daunorubicin
- Phase Ib (decitabine and cedazuridine, venetoclax) (Experimental): Patients receive ASTX727 PO QD on days 1-4 or 1-5 of each cycle and venetoclax PO QD on days 1-28 or days 1-21 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Decitabine and Cedazuridine; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm I (decitabine and cedazuridine, venetoclax); Phase Ib (decitabine and cedazuridine, venetoclax)
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm II (cytarabine, daunorubicin)
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
  Arms: Arm II (cytarabine, daunorubicin)
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
  Arms: Arm I (decitabine and cedazuridine, venetoclax); Phase Ib (decitabine and cedazuridine, venetoclax)
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: Arm I (decitabine and cedazuridine, venetoclax); Phase Ib (decitabine and cedazuridine, venetoclax)

SUMMARY:
This phase Ib/II trial studies the effects of ASTX727 (decitabine and cedazuridine) in combination with venetoclax in treating patients with higher-risk acute myeloid leukemia patients who do not have a change in the gene called fms-like tyrosine kinase 3 (FLT3). Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Cedazuridine is an enzyme inhibitor. It helps to increase the amount of decitabine in the body so that the medication will have a greater effect. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. Venetoclax may stop the growth of cancer cells by blocking BCL-2, a protein needed for cancer cell survival. Venetoclax and decitabine are commonly given together for older patients with AML ASTX727 (a pill form of decitabine + cedazuridine) has been found to be equal to decitabine (given intravenously), and this part of the study is to confirm that venetoclax and ASTX727 is as safe as venetoclax and decitabine given intravenously. This study allows for lowering doses of study drugs to assure the dose chosen for the randomized study (second portion of this trial) is safe and tolerable for people. Giving ASTX727 in combination with venetoclax may help in the treatment of patients with higher-risk acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine and compare the preliminary efficacy of venetoclax +ASTX727 versus (vs.) standard anthracycline induction therapy ('7+3') with a primary endpoint of event-free survival (EFS).

SECONDARY OBJECTIVES:

I. To determine the complete response (complete response [CR] + complete response with incomplete bone marrow recovery [CRi]) rate in patients with treatment naive FLT3 wild type (WT) acute myeloid leukemia (AML) treated with venetoclax and ASTX727 vs. standard anthracycline induction therapy ('7+3').

II. To determine the duration of response (DoR) in patients with treatment naive FLT3WT AML treated with venetoclax and ASTX727 vs. standard anthracycline induction therapy ('7+3').

III. To determine the progression free survival (PFS) of patients with treatment naive FLT3WT AML treated with venetoclax and ASTX727 vs. standard anthracycline induction therapy ('7+3').

IV. To determine the overall response rate (ORR) in patients with treatment naive FLT3WT AML treated with venetoclax and ASTX727 vs. standard anthracycline induction therapy ('7+3').

V. To determine the overall survival (OS) of patients with treatment naive FLT3WT AML treated with venetoclax and ASTX727 vs. standard anthracycline induction therapy ('7+3').

VI. To determine the proportion of patients receiving stem cell transplantation (SCT) in patients with treatment naive FLT3WT AML treated with venetoclax and ASTX727 vs. standard anthracycline induction therapy ('7+3').

VII. To identify mutational burdens in venetoclax +ASTX727 sensitive vs. resistant AML leukemia initiating cells (LICs).

EXPLORATORY OBJECTIVES:

I. To identify transcriptomic signatures in venetoclax +ASTX727 sensitive vs. resistant AML LICs.

II. Determine the utility of high-throughput phenotype-based assessment of drug efficacy for predicting patient response to venetoclax +ASTX727.

III. Determine if treatment failure is a function of therapy sequence or results in resistance to the alternative therapy by conducting a co-clinical trial via patient-derived xenograft (PDX).

IV. To characterize the pharmacokinetics of venetoclax. V. To determine the morphologic leukemia-free state (MLFS) rate in patients with treatment naïve FLT3WT AML treated with venetoclax and ASTX727 vs. 7+3 therapy.

OUTLINE: This is a phase Ib dose de-escalation study followed by a phase II randomized study.

PHASE Ib: Patients receive ASTX727 (decitabine and cedazuridine) orally (PO) once daily (QD) on days 1-4 or 1-5 of each cycle and venetoclax PO QD on days 1-28 or days 1-21 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ASTX727 PO QD at the recommended phase II dose and venetoclax PO QD on days 1-28 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial.

ARM II: Patients receive cytarabine intravenously (IV) over 24 hours on days 1-7 of each cycle and daunorubicin IV over 10-30 minutes on days 1-3 of each cycle. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy throughout the trial.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 18-65 years of age at the time of signing the Informed Consent Form (ICF) and must be able to meet all study requirements. AML patients under the age of 18 are excluded as is being studied in patients under 18 years of age in different venues
* Morphologically confirmed diagnosis of AML in accordance with World Health Organization (WHO) diagnostic criteria
* Adverse risk AML per 2017 European LeukemiaNet (ELN) recommendations
* Subjects must be either treatment naive defined by =< 1 cycle of deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) therapy, no history of cytotoxic chemotherapy for their AML; prior treatment with lenalidomide, hydroxyurea or erythropoiesis-stimulating agents (ESAs) is allowed (prior treatment for myelodysplastic syndrome [MDS] with > 1 cycle of DNMTi is not allowed)
* A bone marrow aspirate and biopsy must be performed, and tissue collected for entrance to the trial
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Recovery to =< grade 1 or baseline of any toxicities due to prior systemic treatments, excluding alopecia
* White blood cell count (WBC) < 25,000 (may be reduced with leukapheresis or hydroxyurea prior to study start)
* Direct bilirubin =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine clearance >= 30 mL/min (per the Cockcroft-Gault formula)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment or have received treatment, they are eligible if they have an undetectable HCV viral load
* Tumor lysis present prior to therapy must be treated accordingly prior to start of therapy
* The effects of venetoclax and ASTX727 on the developing human fetus are unknown. For this reason and because BCL2 inhibitor and DNMTi agents as well as other therapeutic agents used in this trial (cytarabine and daunorubicin) are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal method of birth control or abstinence) prior to study entry and for the duration of study participation, and for 6 months following completion of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception (latex or synthetic condom or abstinence) prior to the study, for the duration of study participation, and 3 months after completion of venetoclax and ASTX727 administration
* Ability to understand and the willingness to sign a written informed consent document
* Adequate cardiac systolic function as measured by ejection fraction (EF) >= 50%

Exclusion Criteria:

* Favorable or intermediate risk AML as defined by 2017 ELN criteria
* Presence of FLT3 TKD or FLT-ITD mutations
* Inability to tolerate oral medication or keep a pill diary
* Active documented central nervous system (CNS) leukemia
* Concurrent treatment with a non-permitted concomitant medication
* Concurrent anticancer treatment, major surgery, or use of any investigational drug within 28 days before the start of trial treatment
* Other malignancy currently being treated or likely to be treated in next 6 months with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ and patients receiving hormonal therapy for prevention of hormone-sensitive cancers
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to venetoclax, ASTX727, or other agents used in study
* Patient must not have received known moderate or strong CYP3A inducers within 7 days of enrollment. Patient must not have known medical conditions requiring chronic therapy of moderate CYP3A inducers. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations (including substance abuse) that would limit compliance with study requirements
* Pregnant women are excluded from this study because venetoclax and ASTX727 have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with venetoclax, breastfeeding should be discontinued if the mother is treated with venetoclax. These potential risks may also apply to other agents used in this study
* Previous exposure to either venetoclax or > 1 cycle of DNMTi (e.g. azacitidine, decitabine, ASTX727, CC486)
* Active, uncontrolled infection as determined by the investigator. Patients with infection under active treatment and controlled with antibiotics are eligible
* Any condition deemed by the investigator to make the patient a poor candidate for clinical trial and/or treatment with investigational agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2026-11-05 (Estimated)

PRIMARY OUTCOMES:
Recommended safe phase 2 dose (RP2D) of decitabine and cedazuridine (ASTX727) in combination with venetoclax (Phase Ib) | End of each cycle (1 cycle = 28 days)
  The highest dose level in which at most 1 patient in 6 experiences dose-limiting toxicity (DLT).
Incidence of adverse events (Phase Ib) | Up to 2 years after completion of study treatment
  Will be tabulated and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Summary statistics will be provided for all adverse events reported. Descriptive statistics, including means, standard deviations, and ranges for continuous parameters, as well as percent and frequencies for categorical parameters, will be presented
Event-free survival (EFS) (Phase II) | Up to 2 years after completion of study treatment
  Will be estimated using the method of Kaplan and Meier and compared among treatments and other important prognostic groups using the log-rank test.

SECONDARY OUTCOMES:
Complete response rate (Phase II) | Up to 2 years after completion of study treatment
  Rate of complete response (CR) + complete response with incomplete bone marrow recovery (CRi).
Duration of response (Phase II) | Up to 2 years after completion of study treatment
  Will be estimated using the method of Kaplan and Meier and compared among treatments and other important prognostic groups using the log-rank test.
Progression-free survival (PFS) (Phase II) | Time from randomization date to the date of progression or death for any reason, assessed up to 2 years after completion of study treatment
  The distribution of PFS will be estimated using the method of Kaplan and Meier. Hazard rate for PFS will be estimated, along with 95% confidence intervals, using the Cox (proportional hazards) regression model.
Overall response rate (Phase II) | Up to 2 years after completion of study treatment
  Rate of partial response (PR) + CRi + CR in patients with treatment naive AML treated with venetoclax and ASTX727.
Overall survival (OS) (Phase II) | Time from randomization to death for any reason, assessed up to 2 years after completion of study treatment
  The distribution of OS will be estimated using the method of Kaplan and Meier. Hazard rate for OS will be estimated, along with 95% confidence intervals, using the Cox (proportional hazards) regression model.
The proportion of treatment naive AML patients receiving stem cell transplantation (SCT) following treatment with venetoclax and ASTX727 (Phase II) | Up to 2 years after completion of study treatment
Mutational burdens in venetoclax + ASTX727 sensitive vs. resistant AML leukemia initiating cells (LICs) (Phase II) | Up to 2 years after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Savona, Principal Investigator — Yale University Cancer Center LAO
Locations (7):
- United States (7):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Yale University, New Haven, Connecticut
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (2):
  • Informed Consent Form: Research Study Informed Consent Document (Phase 2 study) (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT04817241/ICF_000.pdf
  • Informed Consent Form: Research Study Informed Consent Document (Phase 1b) (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT04817241/ICF_001.pdf